CLINICAL TRIAL: NCT01789021
Title: Analytical Performance Evaluation of Blood Glucose Monitoring Systems
Brief Title: Analytical Performance Evaluation of Blood Glucose Monitoring Systems- Investigator Sponsored Contour® XT Comparator Study - Ulm Germany
Acronym: IDT-1206-BA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1206-BA
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: blood glucose monitoring systems; ISO 15197; system accuracy
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Device: 4 blood glucose monitoring systems

SUMMARY:
In this clinical trial, accuracy evaluation of Bayer Contour XT blood glucose monitoring system and blood glucose monitoring systems from other companies across the overall tested glucose range will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Male or female subjects with type 1 or type 2 diabetes or healthy subjects
* For BG adjustment people with type 1 diabetes

Exclusion Criteria:

* Severe acute illness that, in the opinion of the Investigator, might pose additional risk to the patient
* Chronic illness that, in the opinion of the Investigator, might pose additional risk to the patient
* Current condition that, in the opinion of the Investigator, doesn't enable subject to participate in the study
* For BG adjustment people with type 1 diabetes without CHD, condition after myocardial infarction, PAOD, cerebral events or hypoglycaemia unawareness
* Legal incompetence or limited legal competence
* Age < 18 years
* Dependency from the sponsor or the clinical investigator
* Mental incapacity or language barriers precluding adequate compliance with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Differences in accuracy between blood glucose monitoring systems across the overall tested glucose range by comparing the mean absolute value of relative (percent) difference (MARD) between the meter value and the reference value | For each subject, the experimental phase has an expected duration of up to 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Result] Link M, Schmid C, Pleus S, Baumstark A, Rittmeyer D, Haug C, Freckmann G. System Accuracy Evaluation of Four Systems for Self-Monitoring of Blood Glucose Following ISO 15197 Using a Glucose Oxidase and a Hexokinase-Based Comparison Method. J Diabetes Sci Technol. 2015 Apr 14;9(5):1041-50. doi: 10.1177/1932296815580161. PMID 25872967
- [Result] Freckmann G, Pleus S, Link M, Baumstark A, Schmid C, Hogel J, Haug C. Accuracy Evaluation of Four Blood Glucose Monitoring Systems in Unaltered Blood Samples in the Low Glycemic Range and Blood Samples in the Concentration Range Defined by ISO 15197. Diabetes Technol Ther. 2015 Sep;17(9):625-34. doi: 10.1089/dia.2015.0043. Epub 2015 May 19. PMID 26062008